CLINICAL TRIAL: NCT00423410
Title: A First In Man Phase I Study Of EPC2407, A Microtubule Inhibitor Anti-Cancer Drug With Tumor Vascular Endothelial Disrupting Activity: Intravenous Administration Daily For Three Days In Patients With Advanced Solid Tumors And Lymphomas
Brief Title: A Safety Study of EPC2407, A Anti-Cancer Drug With Vascular Disrupting Activity: In Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EpiCept Corporation (Industry)
Responsible Party: Stephane Allard, MD, Chief medical officer, EpiCept
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPC2006-04
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Last update posted 2009-09-10 (Estimated); Status verified 2009-09

CONDITIONS: Advanced Cancer
Keywords: Cancer; Tumor; Lymphoma
MeSH Terms: conditions — Neoplasms; Lymphoma | interventions — crolibulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EPC2407 (crinobulin) (Experimental)
  Interventions: Drug: EPC2407 (crinobulin)

INTERVENTIONS:
Drug: EPC2407 (crinobulin) — IV infusion 1 to 4 hours

SUMMARY:
This study will evaluate the safety, pharmacokinetics (PK), and pharmacodynamic effects of a novel anti-cancer drug, EPC2407, administered to patients with advanced cancer which have not responded to or have recurred following treatment with available therapies

DETAILED DESCRIPTION:
This is a Phase I, open label, multicenter, dose-escalation, safety, pharmacokinetic, and pharmacodynamic study of EPC2407 administered intravenously over 60 minutes on a QDx3 schedule repeated every 21 days. Patients are enrolled and dosed at the level defined by the escalation scheme. The primary goal of the study design is to assess toxicity at the fixed dose levels according to the modified Fibonacci schema.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed solid tumor or lymphoma,which has progressed on standard therapies, for which effective therapy is not available or for patients who are unwilling to undergo such therapies.
2. Males and Females at least 18 years of age
3. Laboratory data as specified below (according to the site's clinical laboratory ranges for normal):

   i. Hematology: ANC >1500 cells/mm3, platelet count >100,000 cells/mm3 and Hemoglobin > 9 gm/L ii. Hepatic: Direct bilirubin <1.5 X ULN; alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 2.5 X ULN. For patients with known liver metastases or liver neoplasms: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 5.0 X ULN iii. Renal: serum creatinine WNL or creatinine clearance >60 mL/min
4. 12-lead electrocardiogram (ECG) QT intervals: QTc ≤ 450 msec for men and ≤ 470 msec for women.
5. Estimated life expectancy of at least 3 months
6. ECOG Performance Status < or = 1
7. Previously treated CNS disease allowed if treatment completed and stable for 4 weeks.
8. For men and women of child-producing potential - willingness to employ appropriate contraceptive methods (including abstinence) during the study
9. Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and to return for the required assessments
10. Cardiac ejection fraction ≥50% by 2D Echocardiogram or > institutional lower limits of normal

Exclusion Criteria:

1. Women who are pregnant or nursing
2. Radiotherapy or any chemotherapy within the previous 21 days or five half lives of prior drug (whichever is shorter). See also exclusion #4 below for patients at risk for cardiac toxicity. Recovery to Grade 1 or less from chemotherapy-induced toxic effect, except alopecia, is required.
3. Major surgery within the last 4 weeks or minor surgery within the last 2 weeks
4. Significant risk of cardiac drug toxicity due to any of the following: a) Active New York Heart Association Class III or IV, b) history of or current congestive heart failure, c) history of myocardial infarction within the last 6 months or ongoing unstable angina, or anthracycline exposure per exclusion #5.
5. Anthracycline exposure exceeding a cumulative dose of 360 mg/m²
6. Known and ongoing HIV, Hepatitis B or Hepatitis C infection
7. Concomitant use of strong inhibitors of the liver microsomal enzymes CYP2C8, CYP2C9, CYP2C19 and CYP3A4.
8. Participation in concurrent study of an investigational agent or device
9. Any other condition including but not limited to major co-morbidities, which in the opinion of the investigator would render the patient ineligible
10. O2 Saturation by pulse oximetry at rest < 90%
11. Concomitant use of drugs that have significant risk of Torsades de Pointes will also be prohibited. Please refer to drugs listed under "Drugs with Risk of Torsades de Pointes"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-12; Primary Completion 2009-04 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Safety | Duration of drug exposure

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Scottsdale Healthcare, Scottsdale, Arizona
  - Tower Oncology Research, Beverly Hills, California
  - Rebecca and John Moores UCSD Cancer Center, San Diego, California